CLINICAL TRIAL: NCT01856972
Title: Does the Addition of Manual Therapy Techniques Increase Gastrocnemius/Soleus Length More Than Stretching Alone?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB13-00096
Record Dates: First submitted 2013-05-14; First posted 2013-05-20 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Muscle Tightness
Keywords: Limited Dorsiflexion Range of Motion; Gastrocnemius tightness; Soleus tightness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Instrument Assisted Soft Tissue Mobilization (Experimental): Subjects randomized into this treatment arm will receive Instrument Assisted Soft Tissue Mobilization to the Gastrocnemius/Soleus complex, as well as a standard stretching/ROM protocol
  Interventions: Procedure: Instrument Assisted Soft Tissue Mobilization; Other: Static stretching/ROM exercises
- Rearfoot joint mobilization (Experimental): Subjects randomized into this treatment arm will receive a rear-foot joint mobilization as well as a standard stretching/ROM protocol
  Interventions: Procedure: Rearfoot joint mobilization; Other: Static stretching/ROM exercises
- Static stretching/ROM exercises (Active Comparator): This is the control group consisting of Static stretching/ROM exercises. No manual intervention is performed with the group. The subjects will perform the standard stretching and ROM protocol
  Interventions: Other: Static stretching/ROM exercises

INTERVENTIONS:
Procedure: Instrument Assisted Soft Tissue Mobilization — IASTM treatment: will be performed with the sound assisted soft tissue mobilization tool #5. Patient will be placed in the prone position with the ankle in a relaxed position. The treating therapist will perform 10 scanning strokes in the caudal, cephalic, medial, lateral directions for a total of 40 strokes over the Gastrocnemius/Soleus complex. The therapist can then perform more concentrated strokes in areas noted by the therapist as tight, with a maximum treatment time of 5 minutes.
  Other Names: IASTM; SASTM
  Arms: Instrument Assisted Soft Tissue Mobilization
Procedure: Rearfoot joint mobilization — A high velocity-low amplitude distractive thrust is directed at the talocrural joint. The procedure is performed with the patient in the supine position. The therapist interlaces hands over the dorsum of the foot with 5th digit placed on talus. The therapist slightly pronates and dorsiflexes the foot. Tension is taken up in a caudal direction until the soft tissue barrier is engaged. A distractive thrust is then applied. This is performed up to 2 times. If the therapist notes a cavitation, the patient is progressed to ROM exercises. If there is no cavitation is noted by the therapist the thrust mobilization is reapplied.
  Other Names: Talocrural caudal thrust mobilization; Talocrural manipulation
  Arms: Rearfoot joint mobilization
Other: Static stretching/ROM exercises — Gastrocnemius stretch at wall 3 sets of 30 second holds. Soleus stretch at wall 3 sets of 30 second holds. Standing bilateral dorsiflexion on step x30 with full ROM. Standing bilateral plantar flexion on step x30 with full ROM.

SUMMARY:
This study will examine the short term effects of adding manual therapy techniques to static stretching in Dorsiflexion (DF) Range of Motion (ROM). The investigators will be studying 2 forms of manual therapy, a rear-foot thrust joint mobilization (TJM), and Instrument assisted soft tissue mobilization (IASTM). By comparing 3 groups: TJM+static stretching versus IASTM + static stretching versus static stretching alone the investigators wish to see if there are any short term benefits in DF ROM by adding either of these interventions to static stretching.

The manual therapy treatment will occur over 2 sessions and DF ROM measurements will be taken 4 times over a 2 week period.

The population that the investigators wish to examine are subjects with healthy feet and ankles, but with limited DF ROM.

The primary objective of this study is to see if subjects with decreased dorsiflexion motion will experience greater increases in dorsiflexion motion with the addition of manual therapy of static stretching alone.

Our hypothesis is subjects who receive manual therapy therapy and static stretching will experience a significant increase in DF ROM as compared to subjects who receive static stretching alone. More specifically subjects who are treated with the IASTM will experience greater results than subjects who are treated with the rear-foot thrust mobilization.

ELIGIBILITY:
Inclusion Criteria:

healthy feet and ankles must have limited dorsiflexion ROM. Limited dorsiflexion will be judged by patient having <12 degrees of DF PROM with knee extended, or <50 degrees of weight bearing DF ROM with the knee flexed.

Exclusion Criteria:

* inability to fully weight bear through their lower extremities
* have <0-90 degrees of ROM in their knees
* inability to follow directions
* presence of a Lower Extremity fracture
* pregnant or nursing

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Weight bearing dorsiflexion Range of Motion | Immediately prior to treatment, Immediately following treatment (same day), 2 day follow up visit,and at 2 weeks (12-16 days after initial session)
  Subjects will perform 3 practice range of motion (ROM) before the first measurement is taken. Subjects will then be measured for Dorsiflexion range of motion with knee in full extension and then with knee flexed 3 times each. With each measurement subjects will be instructed to bend the ankle forward as far as possible without their heel leaving the ground. The average value for these 3 measurements will be calculated and that will be the subjects DF ROM measurement. The change in ROM at each measurement will be the outcome we are measuring

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C Selhorst, MPT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Orthopedic PT East Broad St location, Columbus, Ohio, United States

REFERENCES:
- [Background] Konor MM, Morton S, Eckerson JM, Grindstaff TL. Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2012 Jun;7(3):279-87. PMID 22666642
- [Background] Fong CM, Blackburn JT, Norcross MF, McGrath M, Padua DA. Ankle-dorsiflexion range of motion and landing biomechanics. J Athl Train. 2011 Jan-Feb;46(1):5-10. doi: 10.4085/1062-6050-46.1.5. PMID 21214345
- [Background] Piva SR, Fitzgerald GK, Wisniewski S, Delitto A. Predictors of pain and function outcome after rehabilitation in patients with patellofemoral pain syndrome. J Rehabil Med. 2009 Jul;41(8):604-12. doi: 10.2340/16501977-0372. PMID 19565153
- [Background] Radford JA, Burns J, Buchbinder R, Landorf KB, Cook C. Does stretching increase ankle dorsiflexion range of motion? A systematic review. Br J Sports Med. 2006 Oct;40(10):870-5; discussion 875. doi: 10.1136/bjsm.2006.029348. Epub 2006 Aug 22. PMID 16926259
- [Background] Hammer WI. The effect of mechanical load on degenerated soft tissue. J Bodyw Mov Ther. 2008 Jul;12(3):246-56. doi: 10.1016/j.jbmt.2008.03.007. Epub 2008 Jun 3. PMID 19083680
- [Background] Schaefer JL, Sandrey MA. Effects of a 4-week dynamic-balance-training program supplemented with Graston instrument-assisted soft-tissue mobilization for chronic ankle instability. J Sport Rehabil. 2012 Nov;21(4):313-26. doi: 10.1123/jsr.21.4.313. PMID 23118072
- [Background] Fryer GA, Mudge JM, McLaughlin PA. The effect of talocrural joint manipulation on range of motion at the ankle. J Manipulative Physiol Ther. 2002 Jul-Aug;25(6):384-90. doi: 10.1067/mmt.2002.126129. PMID 12183696
- [Background] Bozymski EM, Isaacs KL. Special diagnostic and therapeutic considerations in elderly patients with upper gastrointestinal disease. J Clin Gastroenterol. 1991;13 Suppl 2:S65-75. doi: 10.1097/00004836-199112002-00009. PMID 1885904